CLINICAL TRIAL: NCT04966702
Title: A Phase III Cluster-randomized, Open-label, Clinical Trial to Study the Safety and Efficacy of Ivermectin Mass Drug Administration to Reduce Malaria Transmission in Two African Settings
Brief Title: Broad One Health Endectocide-based Malaria Intervention in Africa (BOHEMIA)
Acronym: BOHEMIA
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Barcelona Institute for Global Health (Other)
Collaborators: UNITAID (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BOHEMIA
Record Dates: First submitted 2021-06-04; First posted 2021-07-19 (Actual); Last update posted 2025-03-14 (Actual); Status verified 2025-03

CONDITIONS: Malaria
Keywords: ivermectin; malaria; vector control
MeSH Terms: conditions — Malaria | interventions — Albendazole; Ivermectin

STUDY DESIGN:
Intervention Model Description: The BOHEMIA trials are open-label with random assignment to one of 3 treatment arms in Mozambique and 2 in Kenya: (a) ivermectin in humans, (b) ivermectin in humans + livestock (only in Mozambique), or (c) albendazole control.
Masking Description: Open label, assessor-blinded
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Albendazole (Active Comparator): The albendazole group will receive a single dose of 400 mg, given once a month for three months. Generic products will be used in both countries, the final product will be GMP certified and fully bioequivalent with GSK's Albenza®. Bendex (CIPLA) in Mozambique and G-Abzole (Guilin) in Kenya.
  Interventions: Drug: Albendazole Pill
- Ivermectin human (Experimental): The ivermectin group will receive a single dose of 400 mcg/kg, given once a month for three months. Product to be used is Stromectol (Merck) in Mozambique and Ivermectin 3mg USP (Edenbridge) in Kenya.
  Interventions: Drug: Ivermectin Pill
- Ivermectin human and livestock (Mozambique only) (Experimental): The ivermectin group will receive a single dose of 400 mcg/kg, given once a month for three months. Product to be used is Stromectol (Merck). For livestock, locally registered veterinary injectable ivermectin at 1% will be used.
  Interventions: Drug: Ivermectin Pill; Drug: Ivermectin Injectable Product

INTERVENTIONS:
Drug: Albendazole Pill — Using a MDA approach, fieldworkers will administer albendazole using directly observed treatment methodology to participants
  Other Names: Alben, Bendex
  Arms: Albendazole
Drug: Ivermectin Pill — Using a MDA approach, fieldworkers will administer ivermectin using directly observed treatment methodology to participants
  Other Names: Stromectol
  Arms: Ivermectin human; Ivermectin human and livestock (Mozambique only)
Drug: Ivermectin Injectable Product — Veterinary ivermectin injectable will be given to livestock in the relevant cluster
  Other Names: Veterinary Ivermectin 1%
  Arms: Ivermectin human and livestock (Mozambique only)

SUMMARY:
The BOHEMIA program consists of a combination of studies organized around a central community prevention mass drug administration protocol and four sub-studies (i.e.; social science, entomology, health economics, and environmental), each written as an individual protocol. The protocol is central but used in two separate, individually powered trials in Mozambique and Kenya. The trials have been powered on the efficacy outcome and designed to meet the requirements of World Health Organization's (WHO) preferred product characteristics (PPC) for endectocides.

DETAILED DESCRIPTION:
WHO's PPC states that the desired efficacy of an endectocide as stand-alone insecticide in areas of high to moderate transmission is at least 20% reduction in the incidence of clinical malaria (as primary outcome) and incidence of infection (as secondary outcome) in children under 5 years old (the highest incidence age-group in areas with high-transmission), lasting for at least 1 month following a single regimen. Assessing this effect requires a cluster-randomized design with meticulous follow-up of a cohort of children for efficacy and the whole exposed population for safety outcomes, which is the design selected for the BOHEMIA trials.

Two BOHEMIA cluster randomized trials will be carried out in Mozambique (Southern Africa) and Kenya (Eastern Africa). These sites encompass different transmission dynamics that increase the generalizability of results, namely: (a) a gradient of malaria transmission: moderate in Kenya and very high in Mozambique, (b) different species composition of vector population, (c) different rain patterns and environmental conditions, and (d) different livestock species and human/livestock ratios (in Mozambique).

Population:

Co-primary objectives are determined in different populations. Efficacy is primarily determined in a pediatric active cohort (children under 5 years of age in Mozambique and 5-15 years in Kenya), and safety is determined in anyone who receives the drug. Pregnant women and children under 15 kgs are not eligible for treatment.

Treatment Groups:

Two groups of clusters (three in Mozambique) will be randomized to receive (a) ivermectin in humans, (b) ivermectin in humans + livestock (only in Mozambique), or (c) albendazole control. In Mozambique, the study district will be subject to enhanced passive surveillance for malaria.

Primary Outcome Measure:

The primary outcome measure is proposed as incidence in a six-month period given that ivermectin is a short-acting intervention with <1% residual drug at 30 days after each dose. Efficacy assessment will continue 4 months post last dose of ivermectin, and this will include analysis of the vector population. We have proposed the appropriate duration of impact evaluation relevant to the biology of the intervention, and geared towards being able to clean the data, lock the database, and conduct the primary efficacy and safety analysis efficiently.

Estimated Duration of Study:

Throughout the study there will be two different groups of participants enrolled, the ones receiving the treatment (>15 kg) and the ones in the active pediatric cohort for the main outcome of malaria incidence (the ages of highest incidence in each country, under 5 years of age in Mozambique and 5-15 years in Kenya). Each group will participate for different periods of time.

Only the group enrolled in the active pediatric cohort will contribute to the primary efficacy outcome and this group will participate from date of first dose for six months. The group receiving treatment (>15 kg) will contribute to the primary safety outcome and several secondary outcomes (PK, Neglected Tropical Diseases [NTDs]) and this group will participate for four months. Women of child-bearing age will be visited one month after the third dose for a final pregnancy test, any pregnancy occurring during the trial will be followed until birth. The cross-sectional survey will enroll participants of all ages one month after the last Mass Drug Administration (MDA) round.

WHO guidance states that trial design and duration should reflect the nature of the intervention and are left at the discretion of researchers. These trials are robustly powered and are being conducted in moderate to high burden areas, so we believe the risk of failing to find an effect is low and if so, it would throw the utility of the intervention into question.

Advancing the development of this new tool towards implementation in the field can be accomplished in a time frame to contribute to the 2030 Global Technical Strategy (GTS) goals.

ELIGIBILITY:
Inclusion Criteria

For human treatment/safety cohort:

* Residents of the study area
* Male or female weighing more than 15kg
* Adult able to provide written consent
* Minors aged 12 to 17 able to provide assent
* Parent/guardian's able to provide consent for minors
* Negative pregnancy test for women aged between 13 and 49
* Agreement to adhere to study visits and procedures

For pediatric active cohort:

* Children in the age of highest burden at the time of enrollment (under 5 years of age in Mozambique or 5-15 in Kenya)
* Residents of the study area
* Parent/guardian's able to provide consent for minors
* Minors aged 12 to 15 in Kenya able to provide assent

For cross sectionals:

* Residents of the area for at least 3 months prior to enrolment
* Parent/guardian's consent for minors
* Ability to provide assent for minors aged 12 to 17
* Written consent from adults

For livestock treatment:

* Owner/guardian able to provide consent
* Animal expected to spend at least one week every study month inside the cluster border

Exclusion Criteria

For human treatment/safety cohort:

* Known hypersensitivity to ivermectin or albendazole
* Risk of Loa as assessed by travel history to Angola, Cameroon, Chad, Central African Republic, Congo, DR Congo, Equatorial Guinea, Ethiopia, Gabon, Nigeria or Sudan
* Pregnant women
* Lactating women in the first week postpartum
* Children < 15 kg
* Currently participating in another clinical trial
* Unwilling to provide informed consent or assent
* Unwilling to adhere to study visits and/or procedures
* Severely ill either self-reported or in the eyes of the investigator, e.g. defined as need for clinical care, or active or progressive disease interfering with activities of daily living. If in doubt, these criteria can be confirmed after a call with either the site PI/MD/safety officer against a pre-defined list.
* Currently under treatment with inhibitors of CYP3A or P-gp or other drugs that can interfere with the study

For incidence cohort:

* Non-residents
* Currently enrolled in other clinical trial

For cross sectionals:

• Non-residents

For livestock treatment (Mozambique):

* Received ivermectin less than four weeks ago
* Intention to milk or slaughter the animal for human consumption during the withdrawal period (28 days after dosing)
* Calves under 8 weeks and piglets under 6 weeks of age

Ages: 1 Week to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 48145 (Actual)
Dates: Start 2022-03-17 (Actual); Primary Completion 2024-04-15 (Actual); Study Completion 2024-10-03 (Actual)

PRIMARY OUTCOMES:
To determine the safety (in humans) and efficacy of ivermectin MDA, administered to humans, or humans and livestock simultaneously (only in Mozambique) for the prevention of malaria. | 6 months
  Efficacy:
  The efficacy endpoint is primarily measured in children (under 5 years of age in Mozambique and 5-15 years old in Kenya) and safety is determined by anyone who receives the drug.
  Infection incidence in the most vulnerable age group (children under 5 years of age in Mozambique and 5-15 years in Kenya) for 6 months from the moment of the first MDA round in their community. Infection incidence has been chosen as primary endpoint based on the WHOs PPC for endectocides.
To determine the safety (in humans) and efficacy of ivermectin MDA, administered to humans, or humans and livestock simultaneously (only in Mozambique) for the prevention of malaria. | 6 months
  Safety:
  The safety endpoint is determined by anyone who receives the drug.
  Rate of adverse events (AEs) and serious adverse events (SAEs) and difference between ivermectin and albendazole.

SECONDARY OUTCOMES:
To assess the efficacy of the intervention using complementary methods (efficacy). | 6 months
  Time to first positive RDT in children in the cohort.
To assess the efficacy of the intervention using complementary methods (efficacy). | 6 months
  Molecular force of infection in a subset of children in the cohort.
To assess the efficacy of the intervention using complementary methods (efficacy). | 6 months
  Malaria case incidence in all ages presenting at health facility.
To assess the efficacy of the intervention using complementary methods (efficacy). | 6 months
  Malaria prevalence in all ages one month after the last dose.
To assess the efficacy of the intervention using complementary methods (efficacy). | 6 months
  Multiplicity of infection in all ages one month after the last dose.
To assess the safety of the intervention with complementary methods (safety). | 12 months
  Observed tolerability of the dose.
To assess the safety of the intervention with complementary methods (safety). | 12 months
  Rate of Suspected Unexpected Serious Adverse Reactions (SUSARs).
To assess the safety of the intervention with complementary methods (safety). | 12 months
  AEs and SAEs by organ system.
To assess the PK of the proposed ivermectin dose/regime in its relationship with efficacy and safety outcomes (efficacy and safety). | 72 hours
  Whole blood concentrations of ivermectin in dried blood spots.
To assess the impact of ivermectin MDA at the proposed regimen on the prevalence of selected ectoparasitic NTDs (efficacy on NTDs and acceptability). | 6 months
  * Serial prevalence of scabies using a simplified version of the algorithm described by Mahe et al.
  * Serial prevalence of head lice by visual inspection.
  * Serial prevalence of Tunga penetrans via visual inspection of the skin in both feet and applying the Fortaleza scale.
  * Serial prevalence and severity of bed bug infestation by direct questions about bedbugs in the house.
To assess the relationship between malaria incidence in children (under 5 years in Mozambique and 5-15 years in Kenya) and community prevalence at the peak of the malaria season. | 6 months
  Prevalence - incidence correlation:
  - Malaria infection incidence in children (under 5 years in Mozambique and 5-15 years in Kenya) in the pediatric active cohort at community and health facility levels.
To assess the relationship between malaria incidence in children (under 5 years in Mozambique and 5-15 years in Kenya) and community prevalence at the peak of the malaria season. | 6 months
  Prevalence - incidence correlation:
  - Malaria prevalence at all ages.
To assess the relationship between active and passive surveillance for malaria at health facility (only Mozambique). | 18 months
  * Infection incidence in children at community level (active surveillance)
  * Infection incidence in children at health facility level (passive surveillance)
To assess the accuracy for malaria diagnosis of two the different malaria rapid diagnostic tests (RDTs) used in comparison to Polymerase Chain Reaction (PCR) (Mozambique). | 6 months
  Results correlation between HRP2 and pLDH-based RDTs
To assess the accuracy for malaria diagnosis of two the different malaria rapid diagnostic tests (RDTs) used in comparison to PCR (Mozambique). | 6 months
  Results correlation between RDTs and PCR
To assess the accuracy for malaria diagnosis of two the different malaria rapid diagnostic tests (RDTs) used in comparison to PCR (Mozambique). | 6 months
  Proportion of RDT negative but PCR positive infections

OTHER OUTCOMES:
To assess the relationship between self-reported pregnancy status, last menstrual period (LMP), and the results of pregnancy tests in women of reproductive age participating in the study. | 3 months
  To evaluate the correlation between self-reported pregnancy status, the LMP and the results of urine pregnancy tests in women of reproductive age participating in the study
To assess all-cause and malaria-related mortality in intervention and control arms (Mozambique only). | 18 months
  Rate of all-cause and malaria-related mortality as determined by health facility records and BOHEMIA safety reporting during the trial.
To assess all-cause and malaria-related mortality in intervention and control arms (Mozambique only). | 18 months
  Verbal autopsies of deaths of participants on both cohorts (Mozambique).
To estimate the prevalence of relevant CYP and P-gp variations in the target population and subjects suffering from Central Nervous System (CNS)-AEs (Mozambique only). | 3 months
  Case-control association study of ivermectin-associated neurological adverse effects with genetic variation in CYP3A5 and ABCB1 and assess the association of the same genetic variants with ivermectin PK.

CONTACTS AND LOCATIONS:
Overall Officials: Regina Rabinovich, Principal Investigator — Barcelona Institute of Global Health; Carlos Chaccour, Principal Investigator — Barcelona Institute of Global Health
Locations (2):
- KEMRI, Kwale, Kenya
- CISM, Mopeia, Zambezia Province, Mozambique

IPD SHARING:
Plan to Share IPD: Yes
In order to ensure that the Project Results may be shared and ISGlobal will make the fully anonymized data generated by the Project publicly available on open access terms in an appropriate online data repository: (i) at the same time as publication, in relation to data supporting, or which may be necessary to validate, the main findings of any publication; (ii) no later than six (6) months after the end of the Project Term, in relation to all other data which may have public health value
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Protocol and ICF: upon ethical approval SAP: before finishing enrolment CSR and code: within 12 months of completion of the trial
Access Criteria: TBD, Free-to-access, publicly available, searchable institutional website

REFERENCES:
- [Derived] Chaccour C, Nicolas P, Martinho S, Mundaca H, Elobolobo E, Ruiz-Castillo P, Houana A, Montana J, Mbanze J, Casellas A, Macucha A, Mael M, Soares A, Kiuru C, Gutierrez AS, Imputiua S, Constantino L, Vegove V, Cole G, Duthaler U, Ribes M, Mutepa V, Brew J, Munguambe H, Stanulovic S, Xerinda A, Materula F, Gorski N, Wanjiku C, Furnival-Adams J, Tunez L, Sam L, Collins L, Xia K, Hammann F, Rudd M, Rist C, Jones C, Maia M, Candrinho B, Rabinovich NR, Saute F. Ivermectin to reduce malaria transmission- safety and efficacy results from the BOHEMIA cluster randomized trial in Mozambique. EClinicalMedicine. 2025 Nov 7;90:103632. doi: 10.1016/j.eclinm.2025.103632. eCollection 2025 Dec. PMID 41278243
- [Derived] Furnival-Adams J, Houana A, Saute F, Elobolobo E, Rudd M, Nicolas P, Montana J, Martinho S, Mundaca H, Mbanze J, Soares A, Imputiua S, Ruiz-Castillo P, Ribes M, Sanz A, Mamudo Sale M, Macucha A, Casellas A, Lopez V, Vegove V, Mutepa V, Munguambe H, Xerinda A, Materula F, Rabinovich NR, Engelman D, Chaccour C. Direct and indirect protection against scabies through ivermectin mass drug administration designed for malaria in Mozambique: a substudy nested within a cluster-randomised, controlled trial. Lancet Microbe. 2025 Dec;6(12):101189. doi: 10.1016/j.lanmic.2025.101189. Epub 2025 Nov 20. PMID 41274299
- [Derived] Chaccour C, Maia M, Kariuki M, Ruiz-Castillo P, Wanjiku C, Kasiwa L, Brazeal A, Casellas A, Ngama M, Onyango T, Elobolobo E, Kazungu K, Mael M, Wangari W, Nuru K, Otuko R, Sanz A, Ringera I, Matano A, Mitora S, Ribes M, Brew J, Gorski N, Nicolas P, Stanulovic S, Omondi I, Furnival-Adams J, Tunez L, Mbarak J, Vegove V, Yaa E, Mramba S, Kibet Y, Nyambura N, Rotich C, Wanjiru S, Vura M, Wanjiku F, Sam L, Collins L, Xia K, Hammann F, Saute F, Rudd M, Rist C, Jones C, Mwangangi J, Rabinovich NR. Ivermectin to Control Malaria - A Cluster-Randomized Trial. N Engl J Med. 2025 Jul 24;393(4):362-375. doi: 10.1056/NEJMoa2411262. PMID 40700688
- [Derived] Furnival-Adams J, Houana A, Nicolas P, Montana J, Martinho S, Casellas A, Mundaca H, Mbanze J, Soares A, Imputiua S, Ruiz-Castillo P, Ribes M, Sanz A, Sale MM, Macucha A, Elobolobo E, Vegove V, Mutepa V, Munguambe H, Xerinda A, Materula F, Rabinovich R, Saute F, Chaccour C. Collateral benefits of ivermectin mass drug administration designed for malaria against headlice in Mopeia, Mozambique: a cluster randomised controlled trial. Infect Dis Poverty. 2025 Mar 27;14(1):25. doi: 10.1186/s40249-025-01290-z. PMID 40140904
- [Derived] Ruiz-Castillo P, Imputiua S, Xie K, Elobolobo E, Nicolas P, Montana J, Jamisse E, Munguambe H, Materrula F, Casellas A, Deng X, Marathe A, Rabinovich R, Saute F, Chaccour C, Sacoor C. BOHEMIA a cluster randomized trial to assess the impact of an endectocide-based one health approach to malaria in Mozambique: baseline demographics and key malaria indicators. Malar J. 2023 Jun 4;22(1):172. doi: 10.1186/s12936-023-04605-3. PMID 37271818
- [Derived] Chaccour C, Casellas A, Hammann F, Ruiz-Castillo P, Nicolas P, Montana J, Mael M, Selvaraj P, Duthaler U, Mrema S, Kakolwa M, Lyimo I, Okumu F, Marathe A, Schurch R, Elobolobo E, Sacoor C, Saute F, Xia K, Jones C, Rist C, Maia M, Rabinovich NR. BOHEMIA: Broad One Health Endectocide-based Malaria Intervention in Africa-a phase III cluster-randomized, open-label, clinical trial to study the safety and efficacy of ivermectin mass drug administration to reduce malaria transmission in two African settings. Trials. 2023 Feb 21;24(1):128. doi: 10.1186/s13063-023-07098-2. PMID 36810194